CLINICAL TRIAL: NCT00578526
Title: A Randomized, Placebo-controlled Phase II Study to Compare the Efficacy and Safety of SU011248 Versus Placebo in Patients With Advanced Urothelial Transitional Cell Carcinoma Who Have Failed or Are Intolerant to Cisplatin-based Chemotherapy
Brief Title: SU011248 for Platinum-Refractory Urothelial Cancer Evaluation Trial
Acronym: SPRUCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tina Cheng, Principal Investigator, AHS Cancer Control Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPRUCE02
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Urothelial Cancer; Bladder Cancer; Adult
Keywords: urothelial cancer; targeted therapy; antiangiogenesis therapy; SU011248; clinical trial
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): SU011248 - 4 weeks on followed by 2 weeks rest period every 6 weeks
  Interventions: Drug: SU011248
- Arm 2 (Placebo Comparator): 1 50 mg capsule OD PO for 4 weeks with 2 week rest until disease progression. Any patient with disease progression will be unblinded and patients on the placebo arm may then be considered for the open label Sutent treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SU011248 — 50 mg capsule OD PO for 28 days followed by 14 days of rest until tumor progression
  Other Names: Sutent, Sunitinib
  Arms: Arm 1
Drug: Placebo — 50 mg capsule OD PO for 28 days then 14 days rest until disease progression
  Arms: Arm 2

SUMMARY:
The purpose of this study is to find out if SU011248 works and if it is safe in patients with advanced transitional cell carcinoma.

DETAILED DESCRIPTION:
The study objectives include the determination of the antitumor effect of SU011248 in patients with urothelial transitional cell carcinoma and to also determine the toxicities and tolerability of SU011248 in patients with urothelial transitional cell carcinoma who have failed or are intolerant to cisplatin-based chemotherapy.

The primary endpoint of the study is to compare progression free survival at 4 months in patients who received SU011248 plus BSC versus patients who received placebo plus BSC

The secondary endpoint is to compare the objective response rate and duration of response in patients who received SU011248 plus BSC versus patients who received placebo plus BSC, to describe the QOL and safety profile of SU011248 when compared to placebo and to describe the overall survival in patients who received SU011248 plus BSC versus patients who received placebo plus BSC

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven inoperable, metastatic or recurrent transitional cell carcinoma of the urothelial tract
* Mixed histology with predominant TCC allowed.
* Failed, intolerant or ineligible for cisplatin based chemo
* Measurable Disease (RECIST)Not previously irradiated.
* Recovered from previous acute treatment to grade 1(CTCAE Vers. 3.0)
* No weight loss >/- 10% within 28 days of day 0
* Adequate Organ Function

Exclusion Criteria:

* Adenocarcinoma, squamous carcinoma or other histology without any components of transitional carcinoma.
* Small cell histology
* More than one previous systemic chemo
* Excised metastases without remaining measureable disease
* Prior therapy with angiogenesis inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-04; Primary Completion 2014-07-16 (Actual); Study Completion 2014-07-16 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 4 months

SECONDARY OUTCOMES:
objective response rate | Study Duration
duration of response | study duration
Change in health-related quality of life | Study Duration
Number of participants that develop an adverse event to treatment. | Study Duration
Overall Survival | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cheng, M.D., Study Director — Tom Baker Cancer Centre
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario